CLINICAL TRIAL: NCT04703985
Title: Evaluation of the Success of Prophylactic Enteral Nutrition in Therapeutic Intensification With Autograft of Autologous Hematopoietic Cells in Hematology
Acronym: GAGNE
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2019/29
Record Dates: First submitted 2020-12-22; First posted 2021-01-11 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Lymphoma; Myeloma
Keywords: Autologous stem cell transplantation; Enteral feeding; Myeloma; Lymphoma
MeSH Terms: conditions — Lymphoma; Neoplasms, Plasma Cell | interventions — Enteral Nutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients under the protocol of Enteral Nutrition: Patients put under the protocol of Enteral Nutrition adapted to the conditioning autograft (BEAM or Melphalan 200)
  Interventions: Dietary Supplement: Enteral Nutrition

INTERVENTIONS:
Dietary Supplement: Enteral Nutrition — Protocol of Enteral Nutrition adapted to the conditioning autograft (BEAM or Melphalan 200)

SUMMARY:
When the digestive tract is functional, learned societies recommend the use of a nutritional support by enteral feeding. Indeed, it has many advantages (maintenance of gut trophicity, reduction of the risk of infection by reducing the incidence of bacterial translocations,...). It has been used for about fifteen years in hematology departments and offers promising results in the context of allogeneic transplantation with prospective trials in progress (NEPHA study). However, its tolerance has not been studied during autologous transplantation. This study aims to assess the success of enteral nutrition in this setting.

DETAILED DESCRIPTION:
In the literature, there are many studies on the nutritional support to be used during allografts, that highlight the superiority of enteral nutrition over parenteral nutrition in terms of reducing co-morbidities.

Enteral nutrition is the nutritional support recommended by learned societies for therapeutic intensification with autograft of autologous hematopoietic cells in hematology. Nevertheless, enteral nutrition presents difficulties in its implementation and failures (refusal of patients, probes vomiting, neutropenic colitis, etc.), requiring the use of parenteral nutrition in case of failure.

In this context, the study proposes to assess the success and effectiveness of enteral nutrition.

ELIGIBILITY:
Inclusion Criteria:

* Patient with lymphoma or myeloma
* Patient admitted for therapeutic intensification with autologous hematopoietic cells who are eligible for nutritional support by enteral nutrition
* Free, informed and written consent signed by the patient

Exclusion Criteria:

* Refusal of the enteral nutrition
* All patients with absolute or enteral nutrition contraindications:
* Digestive fistula
* Intestinal obstruction
* Intestinal ischemia
* Active digestive bleeding
* Digestive malabsorption (short hail syndrome, bariatric surgery, gastrectomy)
* Trauma to the base of the skull or significant deviation of the nasal septum not allowing the insertion of an naso gastric probe.
* Esophagitis or barrett's esophagus
* Persistent gastro-duodenal dysfunction (gastroparesis)
* Patients admitted for autograft for the treatment of conditions other than lymphoma or myeloma (e. g. solid tumours or leukaemia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lymphoma or myeloma
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2023-11-06 (Actual); Study Completion 2023-11-06 (Actual)

PRIMARY OUTCOMES:
Success rate of enteral feeding | From admission to recovery from aplasia (or transfer to the intensive care unit or death)
  Enteral Nutrition will be considered as a success if : TEI / ER > 70%. On average until recovery from aplasia (or transfer to the intensive care unit or death).
  TEI : Total Energy Intake (per-os + enteral nutrition + glucose solutions) ER : Energy Requirement (assessed patient needs)

SECONDARY OUTCOMES:
Causes of failure of enteral nutrition | From admission to recovery from aplasia (an average of 3 weeks)
  All causes of primary or secondary failure that necessitated the cessation of enteral nutrition
Evolution of total energy intake | Every day from admission to discharge (an average of 4 weeks)
  All sources of energy intake (per-os, enteral nutrition, parenteral nutrition, glucose solutions) These will be compared to the estimated needs of patients and expressed as a % of coverage of these needs
Evolution of albuminemia | Once a week from admission to discharge (an average of 4 weeks)
  Blood test carried out on admission and once a week
Weight evolution | From admission to discharge (an average of 4 weeks)
  Weighing carried out on admission and on discharge. Will be used to calculate the percentage of weight loss and assess nutritional status
Evolution of muscular strength | From admission to discharge (an average of 4 weeks)
  Measurements performed at admission and at discharge of the patient. Muscular strength is measured using a dynamometer (in kg)
Number of bacteremia and type of germs | From admission to discharge (an average of 4 weeks)
Number of transfers to the intensive care unit | From admission to discharge (an average of 4 weeks)
Duration of hospitalization | From admission to discharge (an average of 4 weeks)
  Number of days of hospitalization
Prokinetic and associated antiemetic treatments | From admission to discharge (an average of 4 weeks)
Type conditioning | On admission, between 1 and 7 days before autologous stem cell transplantation
  BEAM or Melphalan 200

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien DAVID, Principal Investigator — University Hospital, Bordeaux
Locations (2):
- France (2):
  - CH de la Côte Basque, Bayonne
  - CHU Bordeaux, Bordeaux

IPD SHARING:
Plan to Share IPD: No